CLINICAL TRIAL: NCT07188636
Title: Development and Validation of the Surgical Mortality Model for Predicting Postoperative Mortality in Non-cardiac Surgery: A Retrospective Multi-center Cohort Study
Brief Title: Prediction of Postoperative Mortality in Patients Undergoing Non-cardiac Surgery: Development and Validation of the Surgical Mortality Model
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Ji-Hoon Sim, Assistant Professor, Asan Medical Center
Other Study IDs: AMC [2022-0755]
Record Dates: First submitted 2025-09-13; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Mortality Prediction
Keywords: surgery; mortality; prediction; model; non cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- Development Cohort: Patients undergoing non-cardiac surgery at Asan Medical Center. This cohort was used to develop the model.
  Interventions: Other: No Intervention: Observational Cohort
- Validation Cohort 1: Patients undergoing non-cardiac surgery at Seoul National University Hospital. This cohort was used for external validation.
  Interventions: Other: No Intervention: Observational Cohort
- Validation Cohort 2: Patients undergoing non-cardiac surgery at Samsung Medical Center. This cohort was also used for external validation.
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — Participants underwent non-cardiac surgery and were followed retrospectively without any experimental intervention. Data were collected from electronic medical records and national death registry to assess postoperative mortality outcomes.

SUMMARY:
This study aims to develop and validate a simple, accurate model to predict mortality after non-cardiac surgery.

DETAILED DESCRIPTION:
This retrospective multi-center cohort study aimed to develop and externally validate a predictive model for postoperative mortality in adult patients undergoing non-cardiac surgery. The development cohort included patients from Asan Medical Center, and validation was performed using data from Seoul National University Hospital and Samsung Medical Center. Mortality was assessed at 30 days, 180 days, 1 year, and overall follow-up. The model was developed using LASSO logistic regression and evaluated for discrimination and calibration across cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older who underwent non-cardiac surgery

Exclusion Criteria:

* Patients who underwent obstetric surgeries
* Transplant donors and recipients
* Patients with incomplete data or missing laboratory values

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing non-cardiac surgery at three tertiary hospitals in South Korea (Asan Medical Center, Seoul National University Hospital, and Samsung Medical Center). Patients with preoperative severe renal dysfunction, kidney transplantation, or missing key variables were excluded. A total of 642,377 patients were included for model development and validation.
Sampling Method: Non-Probability Sample
Enrollment: 642377 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
30-day postoperative mortality | Up to 30 days after surgery
  Death from any cause occurring within 30 days after non-cardiac surgery, ascertained from hospital records and national death registry data.

SECONDARY OUTCOMES:
180-day postoperative mortality | Up to 180 days after surgery
  Death from any cause within 180 days after non-cardiac surgery.
1-year postoperative mortality | Up to 1 year after surgery
  Death from any cause within 365 days after non-cardiac surgery.
Overall postoperative mortality | Through study completion (median follow-up: approximately 5 years, maximum: 13 years)
  Death from any cause during the entire follow-up period after non-cardiac surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Hoon Sim, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No